CLINICAL TRIAL: NCT06805058
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Effect of Comedy Therapy on Pain and Anxiety Levels After Ureterorenoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: okutan4
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Care Acceptor, Health; Pain, Postoperative; Anxiety Postoperative; Surgery
Keywords: comedy therapy; pain; anxiety; surgery
MeSH Terms: conditions — Patient Acceptance of Health Care; Pain, Postoperative; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pre-testpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Comedy therapy (Experimental): After URS surgery, patients whose condition is stable after coming to the clinic will be given a patient introduction form, numerical rating scale, state-trait anxiety scales as a pre-test. Patients will be shown 10-minute Turkish comedy films prepared by the researchers. After the intervention, numerical rating scale, state-trait anxiety scales will be given as a post-test.
  Interventions: Other: comedy therapy
- Control Group (No Intervention): After URS surgery, patients whose condition is stable after coming to the clinic will be given a patient introduction form, numerical rating scale, state-trait anxiety scales as a pre-test. No intervention will be made to control group patients. After a certain waiting period, numerical rating scale, state-trait anxiety scales will be given as a post-test.

INTERVENTIONS:
Other: comedy therapy — Patients will be shown 10-minute Turkish comedy films prepared by the researchers
  Arms: Intervention Group: Comedy therapy

SUMMARY:
The aim is to determine the effect of comedy therapy on pain and anxiety levels in patients after Uretero-Renoscopy (URS) surgery.

The hypotheses of this study; H1-0: Comedy therapy has no effect on pain levels in patients after Uretero-Renoscopy surgery.

H1-1: Comedy therapy has an effect on pain levels in patients after Uretero-Renoscopy surgery.

H2-0: Comedy therapy has no effect on anxiety levels in patients after Uretero-Renoscopy surgery.

H2-1: Comedy therapy has an effect on anxiety levels in patients after Uretero-Renoscopy surgery.

DETAILED DESCRIPTION:
Intervention Group

After URS surgery, patients whose condition is stable after coming to the clinic will be given a patient introduction form, numerical rating scale, state-trait anxiety scales as a pre-test. Patients will be shown 10-minute Turkish comedy films prepared by the researchers. After the intervention, numerical rating scale, state-trait anxiety scales will be given as a post-test.

Control Group

After URS surgery, patients whose condition is stable after coming to the clinic will be given a patient introduction form, numerical rating scale, state-trait anxiety scales as a pre-test. No intervention will be made to control group patients. After a certain waiting period, numerical rating scale, state-trait anxiety scales will be given as a post-test.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Not having any visual or auditory problems,
* Not having any communication problems,
* Not having any psychiatric problems.

Exclusion Criteria:

* Not accepting to participate in the study or wanting to leave,
* Having had complications during the perioperative process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
pain level | It will take approximately 5 minutes
  Patients' pain level will be measured with a "numerical rating scale". In the form, 0 points are evaluated as "no pain", 1-3 points as "mild pain", 4-6 points as "moderate pain", 7 and above points as "severe pain".
anxiety level | It will take approximately 30 minutes
  State and Trait Anxiety Scale:
  The adaptation and arrangement of the scales to Turkish was made by Necla Öner and Le Compte. Both scales consist of 20 items and are graded on a 4-point Likert scale. Scoring is done between 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, Dr., Principal Investigator — Study Principal Investigator Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)